CLINICAL TRIAL: NCT06128031
Title: Psychiatric Assessment of Patients With Anorectal Dyssynergia and the Impact on the Quality of Life
Brief Title: Psychiatric Disorder in Anorectal Dyssynergia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Medhat Hussein, Principal Investigator, Assiut University
Other Study IDs: psycosis&anorectal dyssynergia
Record Dates: First submitted 2023-08-21; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Anorectal Disorder; Psychiatric Disorder
MeSH Terms: conditions — Rectal Diseases; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionaire — Psychiatric interview: this will be assessed by (SCID-5)semi structural clinical interview based on Diagnostic and Statistical manual of Mental disorders-5 criteria
  -Psychometric assessment include; Hamilton depression rating scale(7) and Hamilton anxiety rating scale(8) , used to score the symptoms of anxiety or depression Quality of life assessment: will be assessed by the Patient assessment of constipation-quality of life questionnaire

SUMMARY:
1. evaluate psychiatric disorders among patients with anorectal dyssynergia
2. evaluate the effect of delayed diagnosis of anorectal dyssynergia on the quality of the life

DETAILED DESCRIPTION:
Functional constipation is a functional bowel disorder that presents as persistently difficult, infrequent, or seemingly incomplete defecation.

Subjective and objective definitions of constipation include:

(1) straining, hard stools (hard, inspissated stool), unproductive calls ("want to but cannot"), infrequent stools, or incomplete evacuation. (2) <3 bowel movements per week, daily stool weight <35 g/day, or straining >25% of the time Dyssynergia defecation is common and affects up to one half of patients with chronic constipation. This acquired behavioral problem is due to the inability to coordinate the abdominal and pelvic floor muscles to evacuate stool The etiology of dyssynergic defecation is unclear however it was found that the problem began during childhood in 31% of patients, and after a particular event, such as pregnancy, trauma, or back injury in 29% of patients, and there was no cause in 40% of patients.

The first step in making a diagnosis of dyssynergic defecation is to exclude an underlying metabolic or pathologic disorder .A detailed history, prospective stool diaries, and a careful digital rectal examination will not only identify the nature of bowel dysfunction, but also raise the index of suspicion for this evacuation disorder. Anorectal physiology tests and balloon expulsion test are essential for a diagnosis. Newer techniques such as high-resolution manometry and magnetic resonance defecography can provide mechanistic insights.

. anorectal dyssynergia impact quality of life and cause psychiatric problems such as of anxiety, depression, obsessive compulsiveness, psychoticism, and somatization.

So, the investigators aim to evaluate psychiatric disorders among those patients and impact of delayed diagnosis on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as anorectal dyssynergia with anorectal manometric study

Exclusion Criteria:

* patient with diabetes mellitus ,hypertension ,chronic kidney disease ,and chronic liver disease patients
* patient with neurological disease
* patient with thyroid disease
* patient with past history of psychiatric disorders
* patients with past or current medications or substance induced psychiatric disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all population from 18 years which suffer from chronic conistipation and diagnosed anorectal dyssynergia by rectal manometry or defecogram
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
1-Assess psychiatric disorders among patients with anorectal dyssynergia | through study completion, an average of 1 year
  Review the different types of psychiatric disorders in patients have diagnosed anorectal dyssynergia using SCID-5 ,anxiety and depression Hamilton score (from 0-4,zero refer to no symptoms ,4 refer to sever symptoms ), the summation of them show the type and severity of the condition

SECONDARY OUTCOMES:
The impact of anorectal dyssynergia on the quality of the life | Through study completion, an average of 1 year
  By using survey contain 36 short question about the quality of the life of the patient with anorectal dyssynergia and compare the answer with those of normal people

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa osman, teacher, Study Director — Assiut University

REFERENCES:
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Rao SS, Mudipalli RS, Stessman M, Zimmerman B. Investigation of the utility of colorectal function tests and Rome II criteria in dyssynergic defecation (Anismus). Neurogastroenterol Motil. 2004 Oct;16(5):589-96. doi: 10.1111/j.1365-2982.2004.00526.x. PMID 15500515
- [Background] Rao SS, Tuteja AK, Vellema T, Kempf J, Stessman M. Dyssynergic defecation: demographics, symptoms, stool patterns, and quality of life. J Clin Gastroenterol. 2004 Sep;38(8):680-5. doi: 10.1097/01.mcg.0000135929.78074.8c. PMID 15319652
- [Background] Rao SS, Seaton K, Miller MJ, Schulze K, Brown CK, Paulson J, Zimmerman B. Psychological profiles and quality of life differ between patients with dyssynergia and those with slow transit constipation. J Psychosom Res. 2007 Oct;63(4):441-9. doi: 10.1016/j.jpsychores.2007.05.016. Epub 2007 Aug 1. PMID 17905054
- [Background] Shear MK, Vander Bilt J, Rucci P, Endicott J, Lydiard B, Otto MW, Pollack MH, Chandler L, Williams J, Ali A, Frank DM. Reliability and validity of a structured interview guide for the Hamilton Anxiety Rating Scale (SIGH-A). Depress Anxiety. 2001;13(4):166-78. PMID 11413563
- [Background] Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Arch Gen Psychiatry. 1988 Aug;45(8):742-7. doi: 10.1001/archpsyc.1988.01800320058007. PMID 3395203
- [Background] Hosseinzadeh ST, Poorsaadati S, Radkani B, Forootan M. Psychological disorders in patients with chronic constipation. Gastroenterol Hepatol Bed Bench. 2011 Summer;4(3):159-63. PMID 24834176